CLINICAL TRIAL: NCT00018772
Title: 2779 Epidemiology of Genetic and Acquired Risk Factors for Venous Thrombosis
Brief Title: Risk Factors for Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: HEMA-013-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism
Keywords: coagulation; thrombosis genetic markers
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Deep venous thrombosis is the presence of blood clots, usually in the legs that lead to either local problems or breathing problems if the clot moves to the lungs. This study is designed to assess both clinical conditions as well as common genetic factors that lead to more risk of deep venous thrombosis. Clinical conditions of venous thrombosis include: stroke, malignancy, and situations such as surgery, pregnancy, trauma, or travel.

ELIGIBILITY:
Patients must be 18 years with the ability to understand and consent to questionnaire and blood draw, including understanding of genetic testing..

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 1999-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard Marlar, Ph.D.
Locations (1):
- VAMC, Denver, Colorado, United States